CLINICAL TRIAL: NCT02451891
Title: A Phase Ia Clinical Trial to Assess the Safety and Immunogenicity of MVA-EBO Z Alone and a Heterologous Prime-boost Immunisation With ChAd3-EBO Z and MVA-EBO Z in Healthy UK Volunteers
Brief Title: A Phase I Study to Assess Ebola Vaccines cAd3-EBO Z and MVA-EBO Z
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Long term follow up will take place in a new clinical trial.
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EBL04
Record Dates: First submitted 2015-05-07; First posted 2015-05-22 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2016-08

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

ARMS (5):
- Group 1a (Active Comparator): MVA-EBO Z (1 x 10^8 pfu)
  Interventions: Biological: MVA-EBO Z
- Group 1b (Active Comparator): MVA-EBO Z (1.5 x 10^8 pfu)
  Interventions: Biological: MVA-EBO Z
- Group 2 (Active Comparator): ChAd3-EBO Z (2.5 +/- 1.2 x 10^10 vp) and MVA-EBO Z (1 x 10^8 pfu) after 14 days
  Interventions: Biological: MVA-EBO Z; Biological: ChAd3-EBO Z
- Group 3 (Active Comparator): ChAd3-EBO Z (2.5 +/- 1.2 x 10^10 vp) and MVA-EBO Z (1 x 10^8 pfu) after 28 days
  Interventions: Biological: MVA-EBO Z; Biological: ChAd3-EBO Z
- Group 4 (Active Comparator): ChAd3-EBO Z (2.5 +/- 1.2 x 10^10 vp) and MVA-EBO Z (1.5 x 10^8 pfu) after 28 days
  Interventions: Biological: MVA-EBO Z; Biological: ChAd3-EBO Z

INTERVENTIONS:
Biological: MVA-EBO Z
Biological: ChAd3-EBO Z
  Arms: Group 2; Group 3; Group 4

SUMMARY:
This is a clinical trial in which healthy volunteers will be administered experimental Ebola vaccines. The investigators will vaccinate four groups of volunteers.

Group one will receive the MVA-EBO Z vaccine once at the dose of 1 x 10^8 pfu.

Three groups will receive the prime vaccine cAd3-EBO Z followed by the boost vaccine, MVA EBO Z. The second group of volunteers will receive the boost vaccine after 14 +/-7 days at a dose of 1 x 10^8 pfu and the third and fourth group, after 28 +/- 7 days but at different concentrations of MVA-EBO Z (1 x 10^8 pfu for group 3 and 1.5 x 10^8 pfu for group 4).

The study will assess the safety of the vaccinations, and the immune responses to vaccination. Immune responses are measured by tests on blood samples.

The cAd3-EBO Z and MVA-EBO Z vaccines are called viral vectored vaccines. They are made from viruses which are modified so that they cannot multiply. The viruses have extra DNA in them so that after injection, the body makes Ebola proteins (but Ebola does not develop), so that the immune system builds a response to Ebola without having been infected by it.

Healthy volunteers will be recruited in Oxford and London England. The study will be funded by the Wellcome Trust.

DETAILED DESCRIPTION:
It is important to answer this question to understand how best to deploy the vaccine in an outbreak setting, and to give an indication as to whether booster vaccinations may need to be considered to maintain immunity.

In light of this, the extension study has invited volunteers to attend some further optional follow up visits. It would involve obtaining some further blood tests to look for the same markers of vaccine induced immune response that were looked for in the first part of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years

  * Able and willing (in the Investigator's opinion) to comply with all study requirements
  * Willing to allow the investigators to discuss the volunteer's medical history with their GP
  * For females only, willingness to practice continuous effective contraception (see section 6.3.3) during the study and a negative pregnancy test on the day(s) of screening and vaccination
  * Agreement to refrain from blood donation during the course of the study
  * Provide written informed consent

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational Ebola or Marburg vaccine, a chimpanzee adenovirus, or MVA vectored vaccine or any other investigational vaccine likely to impact on interpretation of the trial data
* Receipt of any live, attenuated vaccine within 28 days prior to enrolment
* Receipt of any subunit or killed vaccine within 14 days prior to enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; functional hyposplenism, recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including urticaria, respiratory difficulty or abdominal pain
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of an anaphylactic reaction
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* History of coeliac disease
* Poorly controlled asthma or thyroid disease
* Seizure in the past 3 years or treatment for seizure disorder in the past 3 years
* Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
* Any other serious chronic illness requiring hospital specialist supervision
* Current anti-tuberculosis prophylaxis or therapy
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Travel to a Ebola or Marburg endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis (see Appendix A)
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the first-in-human administration of MVA-EBO Z alone. This will be done by recording the number of participants who experience adverse events. | 24 weeks
Safety and tolerability of the first-in-human administration of MVA-EBO Z . This will be done by recording the severity of adverse events | 24 weeks
Safety and tolerability of the heterologous prime followed by MVA-EBO Z. This will be done by recording the number of participants who experience adverse events. | 28 weeks
Safety and tolerability of the heterologous prime followed by MVA-EBO Z. This will be done by recording the severity of adverse events | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Venkatraman N, Ndiaye BP, Bowyer G, Wade D, Sridhar S, Wright D, Powlson J, Ndiaye I, Dieye S, Thompson C, Bakhoum M, Morter R, Capone S, Del Sorbo M, Jamieson S, Rampling T, Datoo M, Roberts R, Poulton I, Griffiths O, Ballou WR, Roman F, Lewis DJM, Lawrie A, Imoukhuede E, Gilbert SC, Dieye TN, Ewer KJ, Mboup S, Hill AVS. Safety and Immunogenicity of a Heterologous Prime-Boost Ebola Virus Vaccine Regimen in Healthy Adults in the United Kingdom and Senegal. J Infect Dis. 2019 Apr 8;219(8):1187-1197. doi: 10.1093/infdis/jiy639. PMID 30407513